CLINICAL TRIAL: NCT05131113
Title: Stratification of Patients in Oncogeriatrics and Personalization of Interventions
Acronym: ONKO-FRAIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biogipuzkoa Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ONKO-FRAIL
Record Dates: First submitted 2021-07-29; First posted 2021-11-23 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2023-06

CONDITIONS: Oncology; Solid Tumor, Adult
Keywords: fragility; physical exercise; biomarkers; oncogeriatrics
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group will receive the usual care and hygiene recommendations of the movement
- Interventionist group (Experimental): The interventional group will add an individualized physical exercise program to the usual care.
  Interventions: Other: Physical exercise

INTERVENTIONS:
Other: Physical exercise — Physical exercise
  Arms: Interventionist group

SUMMARY:
Multicenter randomized controlled trial. Patients will be randomly assigned to the control group or the intervention group in each of the health centers.

The control group will receive the usual care, while the intervention group will add an individualized physical exercise program to the usual care.

Cancer is a disease of the elderly. More than 65% of all malignancies affect this population. At the same time, the incidence of cancer cases increases and the need to better understand the biological characteristics of the disease, as well as those of the elderly who suffer from it, is highlighted.

Oncogeriatrics is the area that addresses the care of the elderly patient with cancer, taking into account that physiological aging causes older people to have their own characteristics that require a differential approach in care. The low inclusion in clinical trials of elderly patients and the few specific trials carried out in this subpopulation together with the progressive aging of the population mean that the development of this area has become a priority in health policies.

Therefore, there is a need to focus the research area on supervised physical exercise in older people with cancer in an innovative way, with the aim of generating new hypotheses that overcome existing limitations and facilitate the introduction into the health system of this type of interventions.

DETAILED DESCRIPTION:
It seems useful to have instruments that help to objectively evaluate the fragilty and comorbidity of patients with the intention of adequately indicating the administration of antineoplastic treatment. In addition, nowadays, with the arrival of new less toxic treatments, it is essential to make a good selection of the patients to be treated, since there is a risk of treating patients who are not going to benefit from an active treatment just for having more comfortable medications and with less toxicity.

There are several instruments that can help to better select the patients that the investigators are going to treat and to select the supportive care that can help to better tolerate the proposed treatments while maintaining the best possible quality of life. Some of those instruments are aimed at detecting fragility such as comprehensive geriatric assessment. They identify in more detail the different vulnerabilities that can affect the patient in the benefit vs. toxicity balance of the treatment and in the long-term quality of life

Many authors emphasize the importance of including a physical exercise program during and after cancer treatment. Despite this, older people with cancer usually have low levels of physical activity, and few adhere to the recommendations they receive from health centers. For this reason, involving older people with cancer in a regular physical activity program becomes a challenge for those in charge of health centers.

Some studies have shown that physical exercise can reduce the usual loss of functional capacity and reduce frailty during cancer treatment. On the other hand, physical exercise can help reduce pain, toxicity and improve the completion rate of systemic treatment. Recent studies have found that physical exercise on the days of chemotherapy cycles is safe and may be beneficial in reducing neuropathy and maintaining physical well-being. Additionally, physical exercise can impact one of the most common and strenuous adverse effects of cancer treatment, fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 70 or over.
* Solid cancer.
* Candidates for systemic treatment (chemotherapy, hormone therapy, biological therapies or immunotherapy) if the time that has elapsed since the last dose of treatment has been at least 1 month (washout period).
* Patients with breast, gynecological, lung, pleural, digestive, urological, ENT area, sarcomas, brain tumors, melanomas and patients with tumors of unknown origin will be included.Regarding tumor type and stage for patients with lymphoma: 1) Diffuse large B-cell NHL: include stages I-II if Bulky (>7.5 cm) or R-IPI>1. 2) Hodgkin lymphoma: stages I-II if Bulky (>10 cm). 3) Follicular NHL and marginal NHL without GELF treatment criteria. 4) 80 years old receiving 6 R-mini CHOP cycles.

Exclusion Criteria:

* ECOG ≥3
* cases of advanced dementia
* serious psychiatric illnesses
* Lack of basic fluency in the Basque or Spanish language
* those patients unable to get up from the chair and walk independently with or without auxiliary device.
* Neither will those patients who participate in other studies in which they are undertaking a physical exercise program be included.
* Absolute or relative contraindications in which the risk of adverse effects outweighs the possible benefits such as unstable angina, acute symptomatic heart failure ...

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 186 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-05-03 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery | 12 weeks
  Short Physical Performance Battery (SPPB) evaluates balance, gait ability, and leg strength using a single tool. The score for each part is given in categorical modality (0-4). The best score will be 12 points. 1 point of change in the total score has demostrated to be of clinical relevance.

SECONDARY OUTCOMES:
Integral Geriatric Assessment -Socio-familial situation: | 12 weeks
  Abbreviated Gijón Scale (3-15 pts)
Integral Geriatric Assessment - Basic Activities of Daily Living ( BADL): | 12 weeks
  Barthel Index (0-100 pts)
Integral Geriatric Assessment -Instrumental Activities of Daily Living (IADL): | 12 weeks
  Lawton´s test (0-8 pts)
Integral Geriatric Assessment -Cognitive function: | 12 weeks
  Pfeiffer test (0-10 pts)
Integral Geriatric Assessment - Depression: | 12 weeks
  Yesavage test-short form (0-15 pts) (Yes/No)
Integral Geriatric Assessment -Nutritional status: | 12 weeks
  MNA-SF test (0-14)
Integral Geriatric Assessment -Polypharmacy: | 12 weeks
  Number of chronic drugs consumed by the patient
Integral Geriatric Assessment - Geriatric syndromes: | 12 weeks
  Immobility and pressure ulcers (Yes/No); instability and falls (Yes/No); urinary and faecal incontinence (Yes/No); dementia and acute confusional syndrome ( Yes//No); malnutrition (Yes/No); alterations in sight and hearing (Yes/No);constipation, faecal impaction (Yes/No);depression/insomnia (Yes/No)
Integral Geriatric Assessment -Pain: | 12 weeks
  VAS (0-10 pts)
Integral Geriatric Assessment - Emotional distress: | 12 weeks
  Stress thermometer (0-10 pts)
Cognitive function | 12 weeks
  - Montreal Cognitive Assessment (MOCA) test (0-30 pts)
Anthropometry - Weight: | 12 weeks
  Unit of measure: kg
Anthropometry - Height: | 12 weeks
  Unit of measure: cm
Anthropometry -Waist, hip and calf circumference: | 12 weeks
  Unit of measure: cm
Anthropometry -Blood pressure: | 12 weeks
  - Unit of measure: mmHg
Anthropometry 1: - Bioimpedance (in some centers) 1 | 12 weeks
  · Resistance (Ω)
Anthropometry 2: - Bioimpedance (in some centers) 1 | 12 weeks
  · Phase angle (º)
Biomarkers>> a.1 Inflammation markers (pg/ml or ng/ml): | 12 weeks
  - Interleukins 1beta, 2, 4, 6, and 8 (IL-1 b, IL-2, IL-4, IL-6, and IL-8/CXCL8).
Biomarkers>> a.2 Inflammation markers (pg/ml or ng/ml): | 12 weeks
  - Tumor necrosis factor alpha (TNFa)
Biomarkers>> a.3 Inflammation markers (pg/ml or ng/ml): | 12 weeks
  - Interferon gamma (IFN)
Biomarkers>> a.4 Inflammation markers (pg/ml or ng/ml): | 12 weeks
  - C-reactive protein (CRP)
Biomarkers>> a.5 Inflammation markers (pg/ml or ng/ml): | 12 weeks
  - Brain-derived neurotrophic factor (BDNF)
Biomarkers>> a.6 Inflammation markers (pg/ml or ng/ml): | 12 weeks
  - CMV serology
Biomarkers>> b.1 Endocrine-nutritional and muscle wasting markers (pg/ml or ng/ml): | 12 weeks
  - Insulin-derived growth factor (IGF-1).
Biomarkers>> b.2 Endocrine-nutritional and muscle wasting markers (pg/ml or ng/ml): | 12 weeks
  - Dehydroepiandrosterone sulfate (DHEA sulfate)
Biomarkers>> b.3 Endocrine-nutritional and muscle wasting markers (pg/ml or ng/ml): | 12 weeks
  - Vitamin D
Biomarkers>> b.4 Endocrine-nutritional and muscle wasting markers (pg/ml or ng/ml): | 12 weeks
  - Albumin
Biomarkers>> c. Hematological (AU): | 12 weeks
  Biomarkers in the cell fraction of blood samples. Panel of 7 genes related to aging and frailty in RNA extracted from blood leukocytes, by quantitative PCR (qPCR): EGR1, Hsa-miR454, DDX11L1, G0S2, GJB6, CXCL8 and NSF. This panel has been developed at Biodonostia as a diagnostic and frailty stratification tool (European Patent Application EP3599286).
Functional assessment and frailty: - Steep Ramp test (A) | 12 weeks
  >Heart rate (bpm)
Functional assessment and frailty: - Steep Ramp test (B) | 12 weeks
  >Time spent cycling (min/sec)
Functional assessment and frailty: - Steep Ramp test (C) | 12 weeks
  > Maximum W
Functional assessment and frailty: - Frailty | 12 weeks
  G8 scale ( 0-17); Fried Frailty Phenotype (0-5 pts)
Functional assessment and frailty: - Dynamic balance: | 12 weeks
  8 Foot Up and Go Test (8FUGT) (sec)
Functional assessment and frailty: - Physical activity: 1.Accelerometry | 12 weeks
  Sleep efficiency (%)
Functional assessment and frailty: - Physical activity: 2. Accelerometry | 12 weeks
  Moderate too vigorous physical activity (min/d)
Functional assessment and frailty: - Physical activity: 3. Accelerometry | 12 weeks
  Sedentary time (h/d)
Functional assessment and frailty: - Physical activity: 4. Accelerometry | 12 weeks
  Light physical activity (min/d)
Patient-reported outcomes (PRO): -Fatigue: | 12 weeks
  EORTC QLQ-FA12
Patient-reported outcomes (PRO): - Quality of life: | 12 weeks
  EORTC QLQ-C30
Patient-reported outcomes (PRO): - Nutrition: | 12 weeks
  Simplified Nutritional Appetite Questionnire
Patient-reported outcomes (PRO): - Cognition: | 12 weeks
  Cognitive Failures Questionnaire
Patient-reported outcomes (PRO): - Physical activity: | 12 weeks
  Godin Physical Activity Questionnaire
Adverse events (CTCAE) | 12 weeks
  * Treatment discontinuation (Yes/ No)
  * Dose reduction (Yes/ No)
  * Percentage of treatment completed (Yes/ No)
  * Completion of treatment (Yes/ No)
Factors related to physical exercise adherence | 12 weeks
  Beliefs, barriers, facilitators and self-efficacy in relation to physical exercise ( self-developed questionnaire)
Intervention assessment - Follow-up of the intervention | 12 weeks
  Self- developed questionnaire
Intervention assessment - Adverse events associated with the intervention | 12 weeks
  Self- developed questionnaire
Intervention assessment - Satisfaction with the intervention | 12 weeks
  Self- developed questionnaire

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital Universitario Donostia, San Sebastián, Guipuzcoa
  - Hospital Universitario Basurto, Bilbao
  - Hospital Universitario de Araba, Vitoria-Gasteiz, Álava

REFERENCES:
- [Derived] Garcia-Garcia J, Rodriguez-Larrad A, de Rituerto Zeberio MM, Mediavilla JG, Vicente BL, Artola NT, Etxetxipia IZ, Garmendia I, Alberro A, Otaegui D, Rabasco FB, Caffarel MM, Vrotsou K, Irazusta J, Arrieta H, Pelaez M, Belloso J, Basterretxea L. Effects of a 12-week multicomponent exercise programme on physical function in older adults with cancer: Study protocol for the ONKO-FRAIL randomised controlled trial. J Geriatr Oncol. 2025 Dec 5;17(2):102818. doi: 10.1016/j.jgo.2025.102818. Online ahead of print. PMID 41352214